CLINICAL TRIAL: NCT03877835
Title: Diaphragm-sparing Nerve Blocks for Shoulder Arthroplasty: an Exploratory Feasibility Study
Brief Title: Diaphragm-sparing Nerve Blocks for Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Nordlandssykehuset Bodo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 2018/1934-3
Record Dates: First submitted 2019-02-08; First posted 2019-03-18 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Disease

STUDY DESIGN:
Intervention Model Description: Single intervention
Masking Description: Outcome measures will be performed by an independent assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine (Other): SSNB will be performed with 4 ml ropivacaine 5 mg/ml LSIB will be performed With 15 ml ropivacaine 7.5 mg/ml
  Interventions: Procedure: Peripheral nerve blocks

INTERVENTIONS:
Procedure: Peripheral nerve blocks — LSIB + SSNB

SUMMARY:
The combination of a modified lateral sagittal infraclavicular block and a suprascapular nerve block has not been studied in a cohort of total arthroplasty patients. Such diaphragm-sparing nerve blocks for shoulder arthroplasty may provide a very good anesthetic alternative in lung diseased patients who are in need for total arthroplasty of the shoulder.

DETAILED DESCRIPTION:
The investigators hypothesized that a combination of suprascapular nerve block and lateral sagittal infraclavicular block of the posterior and lateral cords would provide good postoperative analgesia for patients undergoing shoulder arthroplasty.

The primary aims of this study were to document numeric rating scale (NRS, 0-10) and use of morphine equivalents during the first 24 hours after surgery. Secondary aims were to determine the incidence of diaphragm paresis 30 minutes after the block and to quantify postoperative hand grip force at 1 hr.

ELIGIBILITY:
Inclusion Criteria:

* 18-78 years old,
* BMI 20-35 kg.m-2
* ASA physical status 1-3

Exclusion Criteria:

* unable to consent,
* pregnancy,
* pre-existing severe respiratory disease,
* use of anticoagulation drugs other than acetylsalicylic acid or dipyridamol,
* allergy to local anaesthetics,
* patients on regular opioids,
* atrioventricular block,
* peripheral neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
NRS | Postoperatively at 1 hour
  Pain on a 0-10 scale where 0=no pain and 10=unbearable pain
The incidence ipsilateral hemidiaphragmatic paralysis after 30 minutes | 30 minutes after the blocks
  Hemidiaphragmatic paralysis was defined as the absence of diaphragmatic motion during normal respiration, coupled with absent or (paradoxical) cranial diaphragmatic movement when the patient forcefully sniffed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No